CLINICAL TRIAL: NCT07062484
Title: A Real-world Study of the Efficacy and Safety of PD-1 Inhibitors Combined With Chemoradiotherapy in Lung Metastatic Nasopharyngeal Carcinoma
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sichuan Cancer Hospital and Research Institute (Other)
Responsible Party: Principal Investigator, Yangkun Luo, Director, Sichuan Cancer Hospital and Research Institute
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SCCHEC-02-2022-018
Record Dates: First submitted 2025-07-02; First posted 2025-07-14 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-07

CONDITIONS: Lung Metastatic Nasopharyngeal Carcinoma
MeSH Terms: interventions — Cisplatin; Radiotherapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Active Comparator)
  Interventions: Drug: Control: gemcitabine, cisplatin, tirelizumab
- Experimental group (Experimental)
  Interventions: Drug: Experimental: gemcitabine, cisplatin, tirelizumab and radiotherapy

INTERVENTIONS:
Drug: Control: gemcitabine, cisplatin, tirelizumab — PD-1 inhibitors combined with chemotherapy
  Arms: Control Group
Drug: Experimental: gemcitabine, cisplatin, tirelizumab and radiotherapy — PD-1 inhibitors combined with chemoradiotherapy
  Arms: Experimental group

SUMMARY:
This study is a retrospective real-world study. In this study, we plan to collect the clinical data of lung metastatic nasopharyngeal carcinoma patients who received PD-1 inhibitors and chemotherapy combined with or without radiotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. age of at least 18 years;
2. Karnofsky Performance Status (KPS) ≥60;
3. histologically confirmed nasopharyngeal squamous carcinoma;
4. metastatic disease after primary standard treatment (patients who had metastatic diseases over six months after treatment);
5. at least 1 measurable metastatic lesions in lung or mediastinal or pleura (imaging for distant metastases with FDG-PET/CT or chest/abdomen CT with contrast);
6. adequate renal , liver and bone marrow function.

Exclusion Criteria:

1. previous treatment with an immune checkpoint inhibitor;
2. recurrent disease;
3. previous systemic chemotherapy for metastatic disease;
4. symptomatic central nervous system metastases;
5. a history of non-infectious pneumonitis that required glucocorticoids, or active autoimmune disease;
6. severe organ dysfunction or not suitable for chemoradiotherapy;
7. individuals that had serious kidney, heart, blood, nervous system, or liver diseases or psychiatric disorders;
8. individuals that had taken part in any other clinical trials testing other drugs within 3 months of the present study;
9. other patients whom researchers deemed unsuitable to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2025-07 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Objective response rate | 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Sichuan Cancer Hospital and Research Institute, Chengdu, Sichuan, China